CLINICAL TRIAL: NCT06998433
Title: Effect of Platelet-Rich Plasma Versus Placebo in the Treatment of Central Centrifugal Cicatricial Alopecia: A Randomized Clinical Trial
Brief Title: Effect of Platelet-Rich Plasma Versus Placebo in the Treatment of Central Centrifugal Cicatricial Alopecia
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Oyetewa Boluwatito Asempa, Assistant Professor of Dermatology, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-55519
Record Dates: First submitted 2025-04-01; First posted 2025-05-31 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Central Centrifugal Cicatricial Alopecia
Keywords: CCCA; scarring alopecia; alopecia; hair loss; PRP; platelet rich plasma
MeSH Terms: conditions — Alopecia | interventions — Injections; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Study participants and investigators will be blinded to randomization results. The investigators who assess the primary endpoint will be blinded and independent of the investigators who administer the study treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Treatment arm 1 (Experimental): In treatment arm 1, participants will receive a total of three PRP injections spaced four weeks apart (Week 0, Week 4, Week 8).
  Interventions: Biological: Platelet-Rich Plasma (PRP) Injections
- Treatment arm 2 (Experimental): In treatment arm 2, participants will receive a total of four PRP injections; the first three spaced four weeks apart (Week 0, Week 4, Week 8), and a final injection twelve weeks later (Week 20).
  Interventions: Biological: Platelet-Rich Plasma (PRP) Injections
- Placebo arm 1 (Placebo Comparator): In Placebo arm 1, participants will receive a total of three saline injections spaced four weeks apart (Week 0, Week 4, Week 8).
  Interventions: Drug: Saline
- Placebo arm 2 (Placebo Comparator): In placebo arm 2, participants will receive a total of four saline injections; the first three spaced four weeks apart (Week 0, Week 4, Week 8), and a final injection twelve weeks later (Week 20).
  Interventions: Drug: Saline

INTERVENTIONS:
Biological: Platelet-Rich Plasma (PRP) Injections — PRP will be injected into the affected scalp.
  Arms: Treatment arm 1; Treatment arm 2
Drug: Saline — Placebo saline solution will be injected into affected scalp.
  Arms: Placebo arm 1; Placebo arm 2

SUMMARY:
This study aims to investigate whether platelet-rich plasma (PRP) injections can help treat central centrifugal cicatricial alopecia (CCCA), a type of scarring hair loss that mostly affects women of African descent. CCCA is a condition that leads to permanent hair loss, usually starting at the top of the scalp and spreading outward. It can also cause discomfort, such as itching, burning, and pain.

The goal is to see if PRP, which comes from the patient's own blood and is thought to reduce inflammation and promote healing, can stop hair loss and even encourage hair regrowth. PRP has been used to treat other types of hair loss, but it has not been widely studied for CCCA.

Participants in the study will be women of African descent who have been diagnosed with mild to moderate CCCA. Some participants will receive PRP injections, while others will receive a placebo (an inactive treatment) as part of a randomized, double-blind trial. All participants will continue using a topical steroid treatment, which is the standard of care for this condition.

The study will also look at growth factors in participants' blood to understand how they may affect hair loss or regrowth. The goal is to gather information that could lead to better treatments for CCCA, a condition that currently has no standard treatment guidelines.

Although there are risks such as minor discomfort from blood draws and scalp injections and/or a small risk of disease progression, the potential benefits include improved hair growth and a better understanding of CCCA treatments.

DETAILED DESCRIPTION:
Central centrifugal cicatricial alopecia (CCCA) is a common form of permanent hair loss that primarily affects Black women, with up to 20% of this population experiencing the condition. CCCA is characterized by progressive hair loss starting at the crown and spreading outward, often accompanied by symptoms such as burning, itching, and scalp pain. Current treatments focus on reducing inflammation using topical or injectable steroids and oral anti-inflammatory medications. However, these approaches frequently fail to stop hair loss or stimulate hair regrowth, and little is known about the disease's underlying mechanisms. Recent research suggests that CCCA is driven by significant fibrosis out of proportion to the initial inflammation, making it a chronic fibroproliferative disorder that may be similar to conditions like systemic sclerosis, keloids, and uterine fibroids. This scarring complicates treatment and contributes to the physical, emotional, and psychological burden that many Black women with CCCA experience.

Our research proposal aims to evaluate the use of platelet-rich plasma (PRP) injections as a novel therapeutic approach for CCCA. PRP is an autologous treatment in which a patient's blood is processed to concentrate platelets, which contain multiple growth factors and cytokines known to promote tissue regeneration and reduce inflammation and scarring. PRP has been used successfully in other conditions but has not been studied extensively for CCCA. This study will be the first randomized, placebo-controlled trial to assess the efficacy of PRP in treating CCCA in Black women. We hypothesize that PRP's anti-inflammatory and anti-fibrotic properties may slow the progression of the disease and, in some cases, induce hair regrowth. By comparing PRP with placebo injections, we aim to provide conclusive evidence on the treatment's effectiveness.

In addition to evaluating clinical outcomes, we will conduct a secondary experiment to measure growth factor levels in the PRP and platelet-poor plasma of CCCA patients and compare them with levels in women without scarring hair loss. This aspect of the study will provide insight into how specific growth factors may be influencing disease progression or treatment response. By understanding these growth factor profiles, we may be able to predict which patients are more likely to benefit from PRP treatment and potentially refine the approach to enhance its efficacy.

The impact of this study extends beyond CCCA treatment. Our research on growth factor profiles could lead to broader applications in managing other fibrotic skin conditions, such as keloids and systemic sclerosis. This project represents a significant step toward improving hair loss treatments for Black women, providing evidence-based care that takes into account the unique pathophysiology of CCCA. Ultimately, our findings could lead to more personalized treatment strategies, offering hope for improved outcomes and a better quality of life for patients suffering from this challenging condition.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Minimum age of 18 years old
* Self-identification as person of African descent, including African, Afro-Caribbean, Afro-Latino, and/or African American
* Clinical diagnosis of mild to moderate CCCA located on the vertex or fronto-vertex scalp, and as defined by Central Hair Loss Grade stages 1B, 2B, and 3B

Exclusion Criteria:

* Intralesional or systemic anti-inflammatory medications (corticosteroids, tetracycline antibiotics, anti-malarials) or immunosuppressive drugs (cyclosporine, mycophenolate mofetil, methotrexate, azathioprine, janus kinase inhibitors) within 4 weeks of baseline visit
* Pregnant women
* Topical minoxidil, metformin, or retinoic acid for 4 weeks prior to baseline visit
* Severe or end-stage CCCA, Central Hair Loss Grade stage >3B
* Thrombocytopenia (as defined by baseline platelet count < 150,000 platelets per microliter of blood)
* Antiplatelet or platelet altering medications (such as but not limited to aspirin, NSAIDS, clopidogrel, ticagrelor, and prasugrel, cilostazol, and dipyridamole) within 4 weeks of baseline visit
* Diagnosis of other significant concomitant alopecia
* Clinically significant uncontrolled disease, malignancy, or major psychiatric illness requiring hospitalization (as determined by investigator)
* Subjects not willing to follow suggested hair care practices such as limiting/avoiding traction-associated styles

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Physician Global Assessment of Regrowth (PGARG) | At each injection visit: week 0, week 4, week 8, and week 20 (treatment arm 2 and placebo arm 2 only), and three months and six months after final injection
  Physician Global Assessment of Regrowth (PGARG): The average of scores assessed by 2 blinded investigators using comparison of global photography at study end (9 months after initial injection) to photographs from baseline visit. Value of 0 indicates no regrowth; 1, 25% regrowth; 2, 25%-49% regrowth; 3, 50%-74% regrowth; 4, 75%-99% regrowth; 5, 100% regrowth. Average scores between 0.1 and 0.5 will be rounded down to zero. Scores between 0.6 and 0.9 will be rounded up to one.

SECONDARY OUTCOMES:
Change in hair counts | Baseline and three and six months post final treatment.
  Change in hair counts at study end from baseline, including hair density, hair shaft diameter, vellus hair ratio and single hair follicle unit ratio counted digitally using the Canfield Metrix system
Change in Central Hair Loss Grade stage | Baseline and three and six months post final treatment.
  Change in Central Hair Loss Grade stage at study end compared to baseline: Degree of severity of hair loss is graded on a 6-point scale: 0: no hair loss, 1-2: mild hair loss, 3-5: more severe hair loss.
Change in CCCA-QLI | Baseline and three and six months post final treatment.
  Change in CCCA-QLI: Assessment of patients' perception of hair loss and how it relates to their quality of life.
Change in C-CAT | Baseline and three and six months post final treatment.
  Change in C-CAT: Symptom severity questionnaire consisting of numeric ratings of severity of disease progression, pain, pruritus, erythema, and scalp resistance. Values range from 0 (absent) to 2 (moderate-severe) for each symptom. A total score of 0 denotes quiescent disease, less than or equal to 2: mild disease; 3-5: moderate disease; greater than or equal to 6: severe disease activity.
Change in qualitative histological findings at 3 follicular levels | Baseline and six months post final treatment.
Change in quantitative histological findings at 3 follicular levels | Baseline and six months post final treatment.
Change in C-TAS score | Baseline and six months post final treatment
GF levels in plasma and PRP samples of CCCA patients will be compared between responders and non-responders to PRP therapy. | Baseline and six months post final treatment.
Safety evaluations | Baseline and six months post final treatment.
  Safety evaluations, including assessment of adverse events (AEs) such as erythema, worsening pruritus, worsening burning/stinging, scaling, and pain. Investigators will rate AEs as mild, moderate, or severe. Safety evaluations will be compared between treatment and placebo arms.

CONTACTS AND LOCATIONS:
Overall Officials: Oyetewa Asempa, MD, Principal Investigator — Baylor College of Medicine; Assistant Professor of Dermatology, Principal Investigator — Baylor College of Medicine
Locations (1):
- Jamail Specialty Care Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kyei A, Bergfeld WF, Piliang M, Summers P. Medical and environmental risk factors for the development of central centrifugal cicatricial alopecia: a population study. Arch Dermatol. 2011 Aug;147(8):909-14. doi: 10.1001/archdermatol.2011.66. Epub 2011 Apr 11. PMID 21482861
- [Background] Olsen EA, Callender V, McMichael A, Sperling L, Anstrom KJ, Shapiro J, Roberts J, Durden F, Whiting D, Bergfeld W. Central hair loss in African American women: incidence and potential risk factors. J Am Acad Dermatol. 2011 Feb;64(2):245-52. doi: 10.1016/j.jaad.2009.11.693. Epub 2010 Nov 13. PMID 21075478
- [Background] Jackson T, Sow Y, Dinkins J, Aguh C, Omueti Ayoade K, Barbosa V, Burgess C, Callender V, Cotsarelis G, Grimes P, Harvey V, Kindred C, Lester J, Lo Sicco K, Mayo T, McMichael A, Oboite M, Ogunleye T, Olsen E, Osei-Tutu A, Piliang M, Senna M, Shapiro J, Tosti A, Frey C, Adotama P, Taylor SC. Treatment for central centrifugal cicatricial alopecia-Delphi consensus recommendations. J Am Acad Dermatol. 2024 Jun;90(6):1182-1189. doi: 10.1016/j.jaad.2023.12.073. Epub 2024 Feb 9. PMID 38341148
- [Background] Everts P, Onishi K, Jayaram P, Lana JF, Mautner K. Platelet-Rich Plasma: New Performance Understandings and Therapeutic Considerations in 2020. Int J Mol Sci. 2020 Oct 21;21(20):7794. doi: 10.3390/ijms21207794. PMID 33096812